CLINICAL TRIAL: NCT07259590
Title: A Multicenter, Open-Label, Phase Ib/II Clinical Study to Explore the Efficacy, Pharmacokinetics and Safety/Tolerability of GFH375 in Combination With Cetuximab or Chemotherapy in Participants With Advanced Solid Tumors Harboring KRAS G12D Mutation
Brief Title: A Study of GFH375 Combined With Cetuximab or Chemotherapy in Participants With Solid Tumors Harboring KRAS G12D Mutation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFH375X1202
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors Cancer; PDAC; CRC (Colorectal Cancer)
Keywords: solid tumors; KRAS G12D Mutations
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Taxes; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A：GFH375 in combination with Cetuximab (Experimental): Arm A will enroll participants with locally advanced or metastatic solid tumors with KRAS G12D mutation.
  Interventions: Combination Product: GFH375
- Arm B：GFH375 in combination with AG (Experimental): Arm B will enroll participants with locally advanced or metastatic pancreatic ductal adenocarcinoma (PDAC) with KRAS G12D mutation.
  Interventions: Combination Product: GFH375

INTERVENTIONS:
Combination Product: GFH375 — GFH375 once daily (QD) .Cetuximab will be administered via intravenous infusion at a dose of 500 mg/m² every 2 weeks.
  Other Names: Cetuximab
  Arms: Arm A：GFH375 in combination with Cetuximab
Combination Product: GFH375 — GFH375 once daily (QD). Paclitaxel (albumin-bound) at 125 mg/m² and gemcitabine at 1000 mg/m² will be administered via intravenous infusion on Days 1, 8, and 15 of each 4-week cycle.
  Other Names: Paclitaxel (albumin-bound); gemcitabine
  Arms: Arm B：GFH375 in combination with AG

SUMMARY:
This is a Phase Ib/II clinical study aimed at exploring the safety and efficacy of Regimen A (GFH375 in combination with Cetuximab) and Regimen B (GFH375 in combination with AG) in participants with solid tumors.Phase Ib: To evaluate the safety/tolerability and pharmacokinetic (PK) characteristics of GFH375 in combination with cetuximab or AG in participants with solid tumors, and to explore the efficacy of the combination therapy. Phase II: To evaluate the efficacy, safety/tolerability and PK characteristics of the combination therapy, and to explore the correlation between bio-marker and clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the study and sign the informed consent form.
2. Participants receiving Regimen A must be ≥ 18 years old when signing the informed consent form, and participants receiving Arm B must be 18 - 75 years old.
3. Histologically or cytologically confirmed locally advanced unresectable or metastatic solid tumors, with KRAS G12D mutation.
4. Failed standard systemic treatment, or intolerant to standard treatment, or unsuitable for standard treatment, or no standard treatment available.
5. At least one measurable lesions according to RECIST v1.1
6. Participants receiving Regimen A must have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 - 2; participants receiving Regimen B must have an ECOG PS score of 0 - 1.
7. Have sufficient organ function.

Exclusion Criteria:

1. Symptomatic brain metastasis, leptomeningeal metastasis, spinal cord compression, or primary brain tumor.
2. Presence of known coexisting other cancer driver genes.
3. Previous or active history of clinically significant cardiovascular dysfunction.
4. Presence of active infection.
5. History of central nervous system (CNS) diseases.
6. Presence of clinically significant interstitial lung disease, radiation pneumonitis, or immune-related pneumonitis requiring treatment.
7. Newly diagnosed deep vein thrombosis or pulmonary embolism within 3 months before the first administration of the study treatment.
8. Presence of uncontrolled or symptomatic pleural effusion, ascites, or pericardial effusion.
9. Having received major surgery within 28 days before the start of the study treatment; having experienced major trauma within 14 days before the start of the study treatment; or planning to undergo major surgery during the study period.
10. Having received radiotherapy within 4 weeks before the start of the study treatment, or having received palliative radiotherapy for bone metastatic lesions within 2 weeks before the start of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Incidence of Dose-Limiting Toxicity (DLT) Events | up to 28 days
Phase Ib: Incidence and Severity of Adverse Events (AE) and Serious Adverse Events (SAE) | From the first dose until 30 days after the last dose, assessed up to 24 months
Phase II: Objective Response Rate (ORR) Evaluated by RECIST 1.1 | From the first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months

SECONDARY OUTCOMES:
Plasma concentrations of GFH375 | up to 6 months
  Plasma concentrations of GFH375
Phase II: Incidence and Severity of AE and SAE | From the first dose until 30 days after the last dose, assessed up to 24 months
DCR | From the first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  DCR assessed by investigators
TTR | From the first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  TTR assessed by investigators
DOR | From the first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  DoR assessed by investigators
PFS | From the first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1, as Determined by investagors
OS | From the first dose until date of death from any cause, assessed up to 24 months
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No